

IRB Approved: 10/10/2018
IRB Accepted: 11/07/2018
IRB Expiration: 10/09/2019

Title of Study: The Efficacy of Lower Dose Zolpidem for Achieving Satisfactory Sleep in Women with Disordered Sleep

## CONSENT TO CONTACT FOR RESEARCH STUDY

Researchers at Rhode Island Hospital are enrolling adult women in a research study. This study will investigate whether women can get the sleep benefits of Zolpidem (Ambien) on doses lower than 5 mg (the standard available dose) with fewer side effects. Participants will start on very low doses of Zolpidem (0.5mg) and increase the dose by 0.5 mg a day until they achieve satisfactory sleep or the standard prescribed dose for women is reached (5mg), whichever comes first. The study will monitor your quality of sleep and side effects of the lower dose Zolpidem.

If you would like to hear more about this study and would be willing to have a researcher contact you, please sign your name below. A member of the Study Team will contact you to tell you more about the study and answer your questions.

By signing, you understand that you are allowing a researcher at Rhode Island Hospital to contact you to give you more information about the study. This contact does not mean that you are willing to participate in the study. Learning more about the study does not obligate you to sign up for this study.

| YES, a researcher for this | s Study may contact me to tell m | ne more about the study. |
|---|---|---|
| | Signature | Date |
| Printed Name: | | |
| Phone Number: | | |
| Email Address: | | |



| Address 1 (Street | t, Apt Number): | | |
|-------------------|-----------------|---------|---------------|
| Address 2 (City, | State, Zip): | | |
| Best Time to Cor | • / | : | |
| ☐ Morning | Afternoon | Evening | No Preference |